CLINICAL TRIAL: NCT07235553
Title: A Prospective, Multi-center, Randomized, Open-label, Parallel-controlled Non-inferiority Investigation to Evaluate the Efficacy and Safety of the Ultrasonic Surgical System in Clinical Applications
Brief Title: Non-inferiority Investigation to Evaluate the Efficacy and Safety of the Ultrasonic Surgical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Collaborators: Beijing Hospital (Other Government); Peking University Third Hospital (Other); China-Japan Union Hospital, Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US1-080002A
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, randomized, parallel-controlled, non-inferiority study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic Surgical System (Experimental): Ultrasonic Surgical System : ES01; single use shear: SHC23A, SHC36A; handpiece: eHP01
  Interventions: Device: Ultrasonic Surgical System
- HARMONIC System (Active Comparator): HARMONIC System: GEN04; single use shear: ACE23E, ACE36E; handpiece: HP054
  Interventions: Device: HARMONIC System

INTERVENTIONS:
Device: Ultrasonic Surgical System — Generator: ES01; single use shear: SHC23A, SHC36A; handpiece: eHP01
  Arms: Ultrasonic Surgical System
Device: HARMONIC System — Generator: GEN04; single use shear: ACE23E, ACE36E; handpiece: HP054
  Arms: HARMONIC System

SUMMARY:
The objective of this clinical investigation is to evaluate the efficacy and safety of the Ultrasonic Surgical System in the clinical application produced by Ezisurg Medical Co., Ltd.

DETAILED DESCRIPTION:
This clinical investigation is designed as a prospective, multi-center, randomized, parallel-controlled non-inferiority investigation, and the HARMONIC System produced by Ethicon Endo-Surgery, LLC is used as the control product.

Study objective：To evaluate the efficacy and safety of the Ultrasonic Surgical System in the clinical application produced by Ezisurg Medical Co., Ltd.

Target population：Patients who require open or endoscopic surgery using the Ultrasonic Surgical Instruments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily participate in the investigation and sign the Informed Consent Form;
* Male or female subjects aged 18~75;
* Patients who require open or endoscopic surgery using the Ultrasonic Surgical System;
* Those who can communicate well with investigators and comply with investigational requirements.

Exclusion Criteria:

* Patients with severe heart, liver, lung, kidney, brain, blood system diseases, severe metabolic diseases or unable to withstand surgery after systemic assessment;
* Those who with obvious severe local or systemic infection;
* Those who need to undergo the resection of bone tissue and central nervous tissue of the brain and the spinal cord;
* Those who need to undergo contraceptive tubal ligation;
* Those who have a history of alcohol or drug abuse within 6 months before the investigation;
* Women who are pregnant or lactating, or women who plan to become pregnant within 6 months;
* Those who with mental illness;
* Those who have a history of allergies to multiple types of drugs or recent allergic diseases;
* Those who have participated in other clinical investigations in the past 3 months;
* Those who are inappropriate to participate in this clinical investigation for other reasons in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
The overall excellent performance rate | during the surgery
  The overall excellent performance rate will be taken as the primary evaluation indicator. The clinical effect of the investigational product is mainly embodied by its cutting and coagulation functions, and the surgical operators will evaluate the cutting and coagulation functions of the product according to the following criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Wan, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
began enrolling participants beforeJanuary 1, 2019